CLINICAL TRIAL: NCT05896241
Title: EVALUATION OF THE EFFECTIVENESS AND SAFETY OF DOSPRAY® NAZAL SPRAY IN THE SYMPTOMATIC TREATMENT OF PERSISTENT ALLERGIC RHINITIS: A POST-REGISTRATION OBSERVATION STUDY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LeKos LLP (Industry)
Responsible Party: Sponsor
Other Study IDs: № LK-01-D
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients taking Dospray = 63: Patients who were prescribed Dospray as part of routine medical practice
  Interventions: Other: non-interventional study
- Рatients on other alternative treatment = 63: Patients who have been prescribed other alternative treatment as part of routine medical practice
  Interventions: Other: non-interventional study

INTERVENTIONS:
Other: non-interventional study — non-interventional study

SUMMARY:
The combined use of dexamethasone and oxymetazoline has a vasoconstrictive, anti-inflammatory and anti-allergic effect when applied topically in diseases of the upper respiratory tract.

The main goal of this research is Evaluation of the effectiveness of Dospray® nasal spray in the treatment of persistent allergic rhinitis.

The study will involve 126 patients diagnosed with allergic rhinitis:

1. Patients taking Dospray = 63
2. Patients on other alternative treatment = 63 Duration of Patient Participation - 7-10 days (duration of treatment for an individual patient).

DETAILED DESCRIPTION:
Primary task: Overall assessment of the effectiveness of Dospray® nasal spray in the treatment of persistent allergic rhinitis.

Secondary Tasks:

* Symptomatic evaluation of the effectiveness of Dospray® nasal spray in the treatment of persistent allergic rhinitis;
* Evaluation of the effect of Dospray® nasal spray on conjunctive symptoms in the treatment of persistent allergic rhinitis;
* Evaluation of the effect of Dospray® nasal spray on the severity and frequency of nasal symptoms in the treatment of persistent allergic rhinitis;
* Assessment of the quality of life before and after the use of Dospray® nasal spray in the treatment of persistent allergic rhinitis;
* Safety assessment of the use of nasal spray Dospray®.

Study Endpoints:

1. Dynamics of scores on the scale of the reflective Total nasal symptoms score (TNSS) [Time: 7 days]
2. Dynamics of scores on the scale of the individual reflective Total nasal symptoms score (iTNSS) [Time: 7 days]
3. Dynamics of scores on the scale of the reflective Total ocular symptom score (rTOSS)
4. Changes in Visual Analogue Scale (VAS) scores for the severity and frequency of nasal symptoms [Time: 7 days].
5. Dynamics of scores on the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) scores [Time: 7 days]
6. Adverse reactions [Time: 7 days] Number of yellow cards.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 18 to 65 years
* Total TNSS score on the day of inclusion in the study equal to or greater than 4.
* Patients who were prescribed the drug Dospray® or other symptomatic treatment as part of routine medical practice outside the study.
* Voluntary desire to provide informed consent to participate in the study.

Exclusion Criteria:

* Objective symptoms suggestive of renal, hepatic, or heart failure;
* Pregnant and lactating women;
* Patients taking systemic steroids within 30 days prior to inclusion in the study;
* Use of nasal sprays containing corticosteroids within 30 days prior to enrollment in the study;
* Patients receiving immunomodulatory therapy (including Allergen specific immunotherapy (ASIT));
* Patients taking drugs for the treatment of bronchial asthma;
* Patients with polyps in the nasal cavity and / or deformity of the nasal septum requiring surgical correction;
* Infectious diseases of the upper respiratory tract within 14 days before enrollment in the study;
* Patients prone to nosebleeds, having glaucoma, convulsive syndrome or other neuropsychiatric pathologies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons aged ≥18 to 65 years inclusive with a diagnosis of persistent allergic rhinitis who are under outpatient observation.
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Dynamics of scores on the scale of the reflective Total nasal symptoms score (TNSS) | [Time: 7 days]

SECONDARY OUTCOMES:
Dynamics of scores on the scale of the individual reflective Total nasal symptoms score (iTNSS) | [Time: 7 days]
Dynamics of scores on the scale of the reflective Total ocular symptom score (rTOSS) | [Time: 7 days]
Changes in Visual Analogue Scale (VAS) scores for the severity and frequency of nasal symptoms. | [Time: 7 days]
Dynamics of scores on the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) scores | [Time: 7 days]
Adverse reactions - Number of yellow cards. | [Time: 7 days]

CONTACTS AND LOCATIONS:
Locations (2):
- Kazakhstan (2):
  - Allergo Clinic Medical Center, Almaty
  - LLP LOR-Center Ai-Medicus, Almaty

IPD SHARING:
Plan to Share IPD: No